CLINICAL TRIAL: NCT04238234
Title: Comparison of Ultrasound-based Measures of Inferior Vena Cava and Plethysmographic Variability Index for Prediction of Hypotension During Induction of General Anesthesia; Prospective Cohort Study.
Brief Title: IVC Ultrasonography Versus Plethysmographic Variability Index for Prediction of General Anesthesia Induction Hypotension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Other Study IDs: N-68-2021
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Participants will be adult patients (above 18 years), ASA I-II-III, scheduled for elective surgeries under general anesthesia.
  Interventions: Device: IVC Ultrasonography; Device: Plethysmographic variability index (PVI) and perfusion index readings (PI)

INTERVENTIONS:
Device: IVC Ultrasonography — Ultrasound measurements will be performed using a curved transducer set to abdominal mode (1-5 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea). IVC variation will be assessed using ultrasound in the long-axis (sagittal) view. IVC diameter will be measured 1 cm distal to its junction with hepatic vein either by 2-D or M modes via a subcostal approach according to the methodology described by the American Society of Echocardiography . A two-dimensional image of the IVC as it enters the right atrium will be first obtained.
Device: Plethysmographic variability index (PVI) and perfusion index readings (PI) — The PVI and PI will be recorded in the supine position by an anaesthesiologist who was not involved in the further intraoperative monitoring of the patient using Masimo SET ("MightySat 9900, Masimo Corporation, Irvine, CA, USA).
  PVI (%) is a measure of the dynamic change in PI that occurs during one or more complete respiratory cycles, calculated as:
  PVI= [(PImax-PImin)/PImax] x100

SUMMARY:
This thesis aims to evaluate the ability of preoperative plethysmographic variability index to predict post-induction hypotension in comparison with ultrasound measurements of inferior vena cava (IVC) diameter.

DETAILED DESCRIPTION:
Prospective cohort study. Upon arrival to the operating room, routine monitors (ECG, pulse oximetry, and non-invasive blood pressure monitor) will be applied, intravenous line will be secured and routine premedications (ranitidine 50 mg and ondansteron 4mg) will be administrated.

Then inferior vena cava ultrasonography will be performed. Maximum and minimum IVC diameters over a single respiratory cycle will be measured using built-in software. The CI will be calculated as: CI = (dIVCmax - dIVCmin)/dIVCmax , it will be expressed as a percentage.

Plethysmographic variability index and a perfusion index readings will be taken preinduction in the form of three readings on one-minute interval.

Induction of anaesthesia will be achieved using propofol (2 mg/Kg) and atracurium (0.5 mg/Kg). Endotracheal tube will be inserted after 3 minutes of mask ventilation.

Anaesthesia will be maintained by isoflurane (1-1.5%) and atracurium 10 mg increments every 20 minutes. Ringer lactate solution will be infused at a rate of 2 mL/Kg/hour.

Any episode of hypotension (defined as mean arterial pressure < 80% of the baseline reading) will be managed by 5mcg norepinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18years)
* ASA I-II-III
* Patients scheduled for elective surgeries under general anaesthesia.

Exclusion Criteria:

* Operations which will last for less than 15 minutes.
* Patients with cardiac morbidities (impaired contractility with ejection fraction < 40% and tight valvular lesions, unstable angina).
* Patients with heart block and arrhythmia (atrial fibrillation and frequent ventricular or supraventricular premature beat).
* Patient with decompansted respiratory disease (poor functional capacity, generalized wheezes, peripheral O2 saturation < 90% on room air).
* Patients with increased intraabdominal pressure (intrabdominal mass compressing IVC).
* Patients with peripheral vascular disease or long standing DM affecting PVI readings.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be adult patients (above 18 years), ASA I-II-III, scheduled for elective surgeries under general anaesthesia.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the accuracy (Area under receiver operating characteristic curves) of PVI and IVC variation in prediction of post-induction hypotension | 10 minutes before general anesthesia
  Maximum and minimum IVC diameters over a single respiratory cycle will be measured using a built-in software.
  The CI will be calculated as:
  CI = (dIVCmax - dIVCmin)/dIVCmax CI will be expressed as a percentage

SECONDARY OUTCOMES:
Plethysmographic variability index (PVI) and a perfusion index readings (PI) | 3 minutes
  Three readings, on one-minute interval before general anesthesia induction
Maximum and minimum IVC diameters | 10 minutes
  Maximum and minimum IVC diameters over a single respiratory cycle will be measured using built-in software. The CI will be calculated as:
  CI = (dIVCmax - dIVCmin)/dIVCmax , it will be expressed as a percentage.
Mean arterial blood pressure | 20 minutes
  measured at 1-minute intervals starting from the baseline preoperative reading until skin incision as follows: preinduction reading - 1-minute postinduction reading - 2-minute postinduction reading - preintubation reading - one-minute postintubation reading until skin incision
Heart rate | 20 minutes
  measured at 1-minute intervals starting from the baseline preoperative reading until skin incision as follows: preinduction reading - 1-minute postinduction reading - 2-minute postinduction reading - preintubation reading - one-minute postintubation reading until skin incision

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, M.D., Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Kasr alainy, Cairo
  - Almaza Militrary Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Background] Tsuchiya M, Yamada T, Asada A. Pleth variability index predicts hypotension during anesthesia induction. Acta Anaesthesiol Scand. 2010 May;54(5):596-602. doi: 10.1111/j.1399-6576.2010.02225.x. Epub 2010 Mar 10. PMID 20236098